CLINICAL TRIAL: NCT04010357
Title: Targeted Therapy With CDK4/6 Inhibitors in Chemo- Refractory/Relapsed, Rb Wild-type Extensive Small Cell Lung Cancer (SCLC), Large Cell Neuroendocrine Lung Cancer, Extrapulmonary Small Cell Cancers and Other High Grade Neuroendocrine Cancers of the Lung, an Open Label Phase 2 Trial.
Brief Title: Targeted Therapy With CDK4/6 Inhibitors in Chemo-Refractory, Rb Wild-Type Extensive SCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1519
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Small-cell Lung Cancer; Large Cell Neuroendocrine Carcinoma of the Lung; Extrapulmonary Small Cell Carcinoma
Keywords: Platinum refractory disease; Wild Type Rb Extensive Stage SCLC; High grade neuroendocrine cancers of the lung
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Abemaciclib (Experimental): * Subjects will receive Abemaciclib (200 mg), orally every 12 hours on days 1 to 28 of a 28-day cycle for a total of 56 doses per cycle.
  * Subjects will be evaluated after 4 weeks (1st cycle) and then every 8 weeks (2 cycles) with radiographic imaging to assess response to treatment.
  Interventions: Drug: Abemaciclib,

INTERVENTIONS:
Drug: Abemaciclib, — Abemaciclib (CDK4/6 inhibitors) is an investigational drug that works by interrupting the rapid and uncontrolled growth of cancer cells. Some cancer cells develop because their cells overrun the molecular brakes that normally permit cell to divide only when they are needed to replace old ones. These brakes are regulated by a group of enzymes known as cyclin-dependent kinases (CDKs). Alterations causing over-activity of two of these enzymes, CDK4 andCDK6, are found in a variety of cancers, including small cell lung cancer with retinoblastoma (Rb) protein.The drugs work by selectively turning off the overactive CDK4 and CDK6. As a result, the cancer cells' division cycle is halted, preventing them from proliferating.
  Other Names: LY2835219

SUMMARY:
The purpose of this study is to:

* Test how well the study medicine Abemaciclib, a CDK4/6 inhibitor, works to shrink lung cancer tumors in the body.
* Test the safety of Abemaciclib when given to participants with small cell lung cancer (SCLC), large cell neuroendocrine lung cancer, extrapulmonary small cell cancers and other high grade neuroendocrine cancers of the lung. Specifically, this study is looking at SCLC, large cell neuroendocrine lung cancer, extrapulmonary small cell cancers and other high grade neuroendocrine cancers of the lung that have not responded to treatment (refractory) or come back after treatment with chemotherapy (relapsed) as the study medication has been shown to be effective any time the disease relapses not just in the first few months.

DETAILED DESCRIPTION:
This is a multicenter, non-randomized, phase 2, single arm study to determine the efficacy and safety of Abemaciclib as a single agent in patients with biopsy-proven wild type Rb extensive stage of SCLC, with platinum refractory disease (defined as no response after 1-2 cycles of chemotherapy or relapse defined as initial response but relapse after completing platinum-based chemotherapy). Subjects with other tumor types with biopsy proven wild type Rb such as large cell neuroendocrine lung cancer, extrapulmonary small cell cancers and other high grade neuroendocrine cancers of the lung may also be enrolled.

Abemaciclib (CDK4/6 inhibitors) is an investigational drug that works by interrupting the rapid and uncontrolled growth of cancer cells. Some cancer cells develop because their cells overrun the molecular brakes that normally permit cell to divide only when they are needed to replace old ones. These brakes are regulated by a group of enzymes known as cyclin-dependent kinases (CDKs). Alterations causing over-activity of two of these enzymes, CDK4 and CDK6, are found in a variety of cancers, including small cell lung cancer with retinoblastoma (Rb) protein. The drugs work by selectively turning off the overactive CDK4 and CDK6. As a result, the cancer cells' division cycle is halted, preventing them from proliferating.

The objectives of this study include determining:

* Overall Response Rate (ORR) after the first cycle (4 weeks) and then every 8 weeks.
* Progression Free Survival (PFS)assessed at 6 months and Overall Survival (OS).
* Safety and adverse events
* Duration of response in all responders

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically confirmed extensive stage small cell lung cancer, large cell neuroendocrine lung cancer, extrapulmonary small cell cancer or other high grade neuroendocrine cancer of the lung.
* Pathology confirmed Retinoblastoma wild type tested by NGS or ctDNA.
* Subjects must have:
* Platinum refractory disease: defined as no response after 1-2 cycles of chemotherapy, or
* Relapse: defined as initial response but relapse after completing platinum-based chemotherapy.
* Subjects must have measurable disease per the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1.
* Subjects shall have archival tumor material for correlative studies if available. If tissue is not available they still may be eligible for the trial
* Performance status: ECOG Performance status ≤ 2
* Patients who received chemotherapy must have recovered CTCAE Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to enrollment. A washout period of at least 21 days is required between last chemotherapy dose and enrollment (provided the patient did not receive radiotherapy). Please refer to eligibility criteria for specific laboratory requirements.
* Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and enrollment.
* Patients with treated brain metastases are eligible if follow-up brain imaging after CNS-directed therapy shows no evidence of progression.
* The patient is able to swallow oral medications.
* The patient has adequate organ function for all of the following criteria, as defined below:

  * Hematologic system:

    * absolute neutrophil count (ANC) ≥1.5 × 10^9/L
    * Platelets ≥100 × 10^9/L
    * Hemoglobin ≥8g/dL (Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion).
  * Hepatic system:

    * Total bilirubin ≤1.5 × ULN Patients with Gilbert's syndrome with a total bilirubin ≤2.0 times upper limit of normal (ULN) and direct bilirubin within normal limits are permitted.
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 × ULN.
* The effects of the study medication on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (double barrier method of birth control or abstinence) throughout study participation and for 6 months after completing treatment.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior treatment toxicities not resolved to ≤ Grade 1 according to NCI CTCAE Version 5.0 (except alopecia, and neuropathy).
* Subjects receiving any other investigational agents.
* The patient has serious preexisting medical condition(s) that would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* Females who are pregnant or lactating.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Abemaciclib.
* Subjects with uncontrolled intercurrent illness including, syncope of cardiac etiology, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, sudden cardiac arrest, or psychiatric illness/social situations that would limit compliance with study requirements.
* The patient has active bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
* HIV-positive subjects on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Abemaciclib. In addition, these subjects are at increased risk of lethal infections when treated with marrow suppressive therapy. Appropriate studies will be undertaken in subjects receiving combination antiretroviral therapy when indicated.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 2 years from start of study
  Overall Response Rate (ORR) defined as the proportion of subjects in the analysis population who have complete response (CR) or partial response (PR) using RECIST 1.1 criteria at any time during the study. Response for the primary analyses will be determined by independent radiology review.
  CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) according to RECIST 1.1 | At 6 months from start of study
  Defined as the time from allocation to the first documented disease progression according to RECIST 1.1 or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to 10 years from start of study.
  Overall Survival (OS) defined as the time from start of study to death due to any cause.
Safety and adverse events (AE's) and serious adverse events (SAE's) (CTCAE grade version 5.0). | Up to 90 days from end of treatment
  Safety and adverse events (AE's) (CTCAE grade version 5.0) will be assessed by quantifying the toxicities and grades experienced by subjects who have received Abemaciclib (Verzenio®[LY2835219]) including serious adverse events (SAEs). All SE's and grade 3 and 4 AE's will be tabulated.
Duration of response in all responders (DoR using RECIST 1.1) | Up to 2 years from start of study
  Duration of response in all responders (DoR using RECIST 1.1) assessed from the time that measurement criteria met until progressive disease is objectively documented.
  Progressive disease defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Dowlati, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie or influence the results observed from the study.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Investigators who provide a methodologically sound proposal for use of requested data.